CLINICAL TRIAL: NCT05995093
Title: The Proactive Diagnostic Value of Hemostatic Biomarkers in Disseminated Intravascular Coagulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Miao Xu, MD, Principal Investigator, Qilu Hospital of Shandong University
Other Study IDs: Hemostatic Biomarkers in DIC
Record Dates: First submitted 2023-08-06; First posted 2023-08-16 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Disseminated Intravascular Coagulation
Keywords: Thrombosis; Coagulation; Hemostatic Biomarkers; DIC
MeSH Terms: conditions — Disseminated Intravascular Coagulation; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- non-DIC group
  Interventions: Other: no intervention
- pre-DIC group
  Interventions: Other: no intervention
- overt-DIC group
  Interventions: Other: no intervention
- DIC group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University, aiming to evaluate diagnostic performance of hemostatic biomarkers in disseminated intravascular coagulation.

DETAILED DESCRIPTION:
Disseminated intravascular coagulation (DIC) is a life-threatening condition with high mortality, necessitating timely and accurate diagnosis for effective management. However, current diagnostic systems can not recognize DIC at its reversible phase, causing suboptimal treatment outcomes. Consequently, the current diagnostic criteria for DIC lacks earlier laboratory indicators. Therefore, the investigators aimed to assess the diagnostic potential of selected hemostatic biomarkers, including thrombin-antithrombin complex (TAT), soluble thrombomodulin (sTM), tissue plasminogen activator inhibitor complex (tPAI-C), α2-plasmin inhibitor plasmin complex (PIC) and anti-thrombin III (ATIII), in evaluating DIC, allowing for proactive diagnosis before the disease progresses into its irreversible phase.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old, non-perinatal period, a hospitalization length of≥3 days.

Exclusion Criteria:

* primary hematologic diseases, decompensated liver cirrhosis, chemotherapy history.

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients admitted to intensive care unit of Qilu Hospital from 1 January 2021 to 31 December 2022 were involved in our study.
Sampling Method: Probability Sample
Enrollment: 462 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
whether DIC occured | From date of detecting hemostatic biomarkers until the date of first ISTH-DIC scores ≥5, assessed up to 7 days.
  DIC includes pre-DIC and overt-DIC

SECONDARY OUTCOMES:
whether death occurred | From date of admission until the date of death, assessed up to 5 months
  Based on the death records in the electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Miao Xu, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Miao Xu, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: No